CLINICAL TRIAL: NCT07071896
Title: Strong Survivors: A Prospective Study of Video-assisted Exercise Program for the Breast Cancer Survivors
Brief Title: A Prospective Study of Video-assisted Exercise Program for the Breast Cancer Survivors
Acronym: StrongSurvivor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Sara Grossi, Assistant Professor of Clinical Surgery, Breast Surgical Oncology, University of California San Diego Comprehensive Breast Health Center, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 809843
Record Dates: First submitted 2025-03-26; First posted 2025-07-17 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Mastectomy
Keywords: Exercise, Mastectomy; rehabilitation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Strong Survivors (Experimental): 16 week, twice weekly, remote exercise program
  Interventions: Other: 16 weeks remotely exercise program

INTERVENTIONS:
Other: 16 weeks remotely exercise program — 16 weeks, twice per week, remotely exercise program

SUMMARY:
The investigators cancer rehabilitation/recovery program, Strong Survivor, has been designed to be delivered digitally, and while there are many such programs currently available on the internet, especially in the time of COVID-19, the novel feature of this program is the delivery of semi-individualized instruction in real time within a small group setting. The program was designed with physician input and by exercise physiologists and a Doctor of Physical Therapy candidate, all with extensive training in both group and individualized exercise for geriatric and cancer survivor populations. Strong Survivor is 16-week iterative curricular program with three core components: aerobic fitness, balance and mobility, and muscular strength and power. Classes will be held twice per week. The first 4 classes will be deployed in a small class of up to 5 people (first 2 weeks), then one class per week with the small class and one class per week is with a larger class of up to 15 people (weeks 3 and 4). The program is then continued for 12 additional weeks in a larger class using principles and exercises specifically trained during the small group classes.

All the exercises offered over the course of the intervention are appropriate for the target population and are standardized so all participants receive the same basic instruction, but level of difficulty is scaled to participant experience, capability, and musculoskeletal limitations.

Participants will need to have a minimal adequate space and technology to accommodate this instructional method. Specifically, they will require an internet connected device with a camera that is at least 7 inches square. (tablet size or larger).

Additionally, participants' will need to have adequate space to both set up a computer/camera and move around. The minimal acceptable space for this is 6+ feet with an unobstructed view (from a table for instance) of a 2 x 2 open space.

All study participants will complete a clinic visit before they join the classes and after the last class to evaluate cardiorespiratory fitness, strength, balance and posture and answer questionnaires about quality of life and system usability.

DETAILED DESCRIPTION:
Recovery Following Surgery Program: The investigators cancer recovery program, Strong Survivors is designed to be delivered digitally, and while there are many such programs currently available on the internet, especially in the time of COVID-19, the novel feature of this program is the delivery of semi-individualized instruction in real time within a small group setting.

The program was designed with physician input and by exercise physiologists and a Doctor of Physical Therapy, all with extensive training in both group and individualized exercise for geriatric populations, and with the input of individuals with experience working with cancer survivors. As such, Strong Survivors is a 16-week iterative curricular program with three core components: cardiovascular fitness, balance and postural stability, and muscular strength and power. All the exercises offered over the course of the intervention are appropriate for the target population and are standardized so all participants receive the same basic instruction, but level of difficulty is scaled to participant experience, capability, and musculoskeletal limitations.

Participants will need to have a minimal adequate space and technology to accommodate this instructional method. Specifically, they will require an internet connected device with a camera that is at least 7 inches square. (tablet size or larger). While a cell phone is likely adequate for the investigators to see participants, it is not sufficiently large for them to see and follow exercise instruction.

Additionally, participants will need to have adequate space to both set up a computer/camera and move around. The minimal acceptable space for this is 6+ feet with an unobstructed view (from a table for instance) of a 2 x 2 open space. Participants will be coached to place the computer/camera/tablet/etc. at the position ~6 feet away and then stay within the 2x2 foot viewing area during exercise during the at-home zoom based testing (that occurs before the exercise sessions begin) Participants will be recruited so that they begin instruction in groups of 5 (i.e. the intervention will start as soon as 5 participants are recruited) and provided with 2 classes per week for 2 weeks where fundamental exercises are trained and reviewed. The following 2 weeks participants will continue to receive 1 small group class and will also be "added" to the large group class for 1 class per week. For the remaining three months of the intervention (12 weeks) participants will continue to engage in 2 large group classes per week.

Small group classes will be organized at the time of recruitment at 2x per week that matches the scheduling needs of all participants. This will, necessarily, be different for each recruited cohort.

Small group instruction: Five (5) participants will be paired with a master trainer (i.e. >1 year experience training in the zoom based environment and MS degree in exercise physiology, kinesiology, or athletic training) and a junior assistant. The master trainer will provide instruction and review participant performance while the junior assistant will provide support in terms of ensuring appropriate camera positioning (both for instructor and participant) and participant observation for signs of undue distress or difficulty.

Larger group instruction: After 2 weeks of small group instruction participants will be added to the growing group of individuals who have completed the small group instruction but not an additional 12 weeks. In concept this group could grow to infinite levels, but for the purposes of substudy 1 the largest the group could ever be is 15 individuals (the entire cohort). The larger group will also have a master trainer (i.e. >1 year experience training in the zoom based environment and MS degree in exercise physiology, kinesiology, or athletic training) and a junior assistant but will also be joined by a second junior trainer (BS or higher in exercise physiology, kinesiology, or athletic training or certification by a national recognized organization for personal training like ACSM, NASM, or ACE). One of the trainers will always be specifically monitoring participants to provide cues to ensure safety and maximize exercise benefits. The other trainer will both model exercises and provide feedback and the junior assistant will provide support in terms of ensuring appropriate camera positioning and providing participant observation.

All study participants will complete a clinic visit before they join the classes and after the last class to evaluate cardiorespiratory fitness, strength, balance and posture and answer questionnaires about quality of life and system usability.

ELIGIBILITY:
In order to be eligible to participate in this study, an individual must meet all the following criteria:

1. Persons, aged 18+
2. Undergone breast cancer surgery within the 4 weeks of being contacted for pre-screening

   a. Acceptable surgery includes unilateral or bilateral mastectomy (Lymph node surgery is NOT required but is still acceptable)
3. Own a computer or alternative device capable of real-time Zoom videoconferencing, including access to internet or cellular connectivity sufficient in broadband. This requires a screen of at least 7 inches (a cell phone is large enough for us to see the participant, but not for the participant to see us).
4. Provision of signed and dated informed consent form
5. Stated willingness to comply with all study procedures and availability for the duration of the study

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Have sustained a previous fall-related fracture within the last 2 years;
2. have poorly controlled cardiovascular disease, pulmonary disease, or a debilitating musculoskeletal or neurological condition severely limiting function/ability to perform the exercise program as determined by the breast surgeon at screening for trial enrollment
3. experience vertigo or dizziness/light headedness observed at enrollment or during initial occupational therapy evaluation.
4. are on multiple benzodiazepine or neuroleptic medications.
5. Pregnant or trying to become pregnant

   -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-23 (Estimated)

PRIMARY OUTCOMES:
Attendance | 16 weeks
  The number of sessions each participant attended (out of the total number of sessions offered) will be recorded and used to evaluate engagement in the tele-video real time exercise program in a geriatric breast cancer patient population.
  A participant is considered to have completed the study if he or she has completed all phases of the study including responding to follow up queries regarding falls for up to 1 year following the final measurement visit. Acceptability is based on attendance.

SECONDARY OUTCOMES:
Cardiorespiratory Fitness: Time taken to reach 85% of age predicted heart rate max | Before the beginning and at the end of the 16 weeks program
  The time taken to reach 85% of age predicted heart rate max , from a submaximal exercise testing on a treadmill, will be used to evaluate Cardiorespiratory Fitness; pre and post program times will be compared for each study participant.
Strength and Balance | Before the beginning and at the end of the 16 weeks program
  Short Physical Performance Battery test (4-part validated scale for fall risk) will be used to evaluate Strength and Balance
Fall Risk assessment | Before the beginning and at the end of the 16 weeks program
  The Timed Up and Go, Standardized assessment of functional mobility, will be used for Fall Risk assessment
Balance | Before the beginning and at the end of the 16 weeks program
  The Better Balance Testing, measure of proprioceptive and vestibular function utilizing computerized dynamic posturography, will be use to measure balance
Fall Risk | Before the beginning and at the end of the 16 weeks program
  The 25 foot walk, standardized assessment of gait speed and variability associated with fall risk, will be used to evaluate fall risk
Muscular Strength | Before the beginning and at the end of the 16 weeks program
  The 30 Second Chair Stands, common field measure of muscular strength and endurance of the legs, will be used to evaluate legs muscular strength. This score is evaluated relative to a person's age and gender and a lower score in seconds indicates a shorter time to complete the task and represents higher strength and endurance of legs.
Posture | Before the beginning and at the end of the 16 weeks program
  The Occipital to Wall Distance, measurement of kyphotic curvature of the spine, will be used to assess posture
Posture | Before the beginning and at the end of the 16 weeks program
  The Block Measurement, measurement of kyphotic curvature of the spine, will be used to assess posture
Posture | Before the beginning and at the end of the 16 weeks program
  Multiple measures of height, while standing normally versus standing "as tall as possible" (indicative of non-specific postural deficiencies) will be used to evaluate posture
Body Composition | Before the beginning and at the end of the 16 weeks program
  Bio-electrical Impedance, non-invasive assessment of body composition, will be used to evaluate fat mass and muscle mass; those will be measured at the beginning of the program and the end of the program and the difference will be calculated for each study participant. Bioimpedance data can estimate parameters like body fat, lean body mass, and total body water which are calculated as percentages. While height and weight data are gathered during the bioimpedance measurement, they are not a specific reportable outcome measure.
Physical Activity level | Before the beginning and at the end of the 16 weeks program
  Accelerometry, non Invasive home based measure of activity, will be used to evaluate the time spent in moderate-to-vigorous physical activity (MVPA) before the program and at the end of the program; the difference in time spent in MVPA will be calculated for each study participant. The accelerometer will be worn for a week before the program begins and for a week after the program.
Quality of Life assessment via PROMIS-29 questionnaire | Before the beginning and at the end of the 16 weeks program
  The PROMIS-29 questionnaire is a patient-reported outcome (PRO) measure that assesses seven key health domains to evaluate Physical Function, Fatigue, Pain Interference, Depression, Anxiety, Ability to Participate in Social Roles and Activities, Sleep Disturbance and Pain Intensity. Raw scores range from 4 to 20 in each domain with the lowest score of 4 indicating no issues and maximum 20 most issues. It is scored by averaging all item responses for each dimension to create subscores, which are then combined to produce global physical and mental health scores. The pain scale is just one question with zero having no pain to 10 being worst pain. Changes in score from before the program to after the program will be calculated for each study participant.
System Usability | At the end of the 16 weeks program
  System Usability Scale (SUS) is a validated questionnaire designed to understand the ease of use of new systems or programs using a 5 element Likert scale per question. A higher score indicates a higher acceptability. SUS will be administered at the end of the program.
Quality of life using FACT B questionnaire | Before the beginning and at the end of the 16 weeks program
  The Functional Assessment of Cancer Therapy - Breast (FACT-B) is a 37-item instrument designed to measure five domains of Health-Related Quality of Life in breast cancer patients: Physical (PWB), social (SWB), emotional (EWB), functional well-being (FWB) as well as a breast-cancer subscale (BCS). Questions ask about the last 7 days and responses are on a 5 point Likert-type scale. Multiplying the sum of the item scores by the number of items in the subscale, then dividing by the number of items answered produces a subscale score (from 0 to 28 for PWB, SWB, FWB; 0 to 24 for EWB; 0 to 40 for BCS). Adding subscale scores will derive total scores. The higher the score, the better the Quality of Life. Scores will be calculated for each participant and before and after program scores will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD, San Diego, California, United States